CLINICAL TRIAL: NCT02020811
Title: A Study to Assess the Functionality of Pro-IV's IMMAGES Infusion System in Patients Hospitalized in Bait Balev, Receiving Intravenous Therapy
Brief Title: Safety and Efficacy of Immages System in Patients Recieving IV Therapy
Acronym: IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PRo-IV (Industry)
Collaborators: Bait Balev Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BBALEV-1
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-05

CONDITIONS: Sepsis; Bacteriemia; CHF
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sentinel arm (Experimental): all patients will be recieving Iv therapy by using the sentinel controller, a device that is mounted on the IV administration set.
  Interventions: Device: Sentinel

INTERVENTIONS:
Device: Sentinel

SUMMARY:
The study will evaluate the functionality of IMMAGES , an intravenous infusion device system, in patients hospitalized in Bait Balev hospital. The study will aim to determine how the IMMAGES system integrates within IV infusion therapy regime and what are the advantages and disadvantages, if any, of using this system within the prescribed setting.

DETAILED DESCRIPTION:
Using the IMMAGES system in patients recieving IV therapy will provide the nursing teams on-line information regarding the infusions and will allow them to monitor and manage the treatments in real-time, providing better and safer care for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Patients requiring infusion therapy
  2. Patients receiving infusion therapy by gravity flow or by pump
  3. patients are scheduled to receive at least once a day an infusion therapy
  4. Patients are scheduled to receive an infusion therapy for at least 3 days
  5. Adult over age of 18 years
  6. Informed consent form signed by patient.

     Exclusion Criteria:

  <!-- -->

  1. Informed consent form not signed
  2. Patients are scheduled to receive less than once a day an infusion therapy
  3. patients to receive less than 3 days of infusion therapy
  4. patients not hospitalized in a ward that is participating in the study.
  5. patients participating in another clinical study or clinical field test
  6. Patients require isolation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Successful operation of IMMAGES defined by patient receiving the prescribed IV medication using the IMMAGES system , openning of the controller valve including using the smartphone application and the management software | as long as the patient is reciving the IV prescribed medication, and no longer than 10 days

SECONDARY OUTCOMES:
- Detection of medical errors by IMMAGES | up to 5 minutes from activating the controller on the IV line
  If there is an error related to administration of wrong drug. to the wrong patient , on the wrong timing - the valve of the controller will not open , and the IV line will stay closed, and the patient will not get the wrong drug.

CONTACTS AND LOCATIONS:
Overall Officials: michal devir, MD, Study Chair — PRo-IV
Locations (1):
- Bait Balev hospital, Bat Yam, Israel